CLINICAL TRIAL: NCT07306832
Title: A Phase 1b Study of the Safety and Pharmacokinetics of Pivekimab Sunirine in Pediatric Subjects With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Study to Assess Adverse Events and How Intravenous (IV) Pivekimab Sunirine Moves Through the Body in Pediatric Participants With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-692; 2024-520125-36 (Other: EU CT)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Relapsed; Refractory; Pivekimab Sunirine; PVEK; Pediatric
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: Pivekimab Sunirine Ages 2 to < 6 Years (Experimental): Participants will receive pivekimab sunirine, as part of the approximately 28 month study duration. If enrolled, subjects aged 6 months to less than 2 years will be included in Cohort 1
  Interventions: Drug: Pivekimab Sunirine
- Cohort 2: Pivekimab Sunirine Ages 6 to < 12 Years (Experimental): Participants will receive pivekimab sunirine, as part of the approximately 28 month study duration.
  Interventions: Drug: Pivekimab Sunirine
- Cohort 3: Pivekimab Sunirine Ages 12 to < 17 Years (Experimental): Participants will receive pivekimab sunirine, as part of the approximately 28 month study duration.
  Interventions: Drug: Pivekimab Sunirine

INTERVENTIONS:
Drug: Pivekimab Sunirine — Intravenous

SUMMARY:
Acute myeloid leukemia (AML) is an aggressive blood cancer, withwith few options for participants who relapse after treatment or who don't respond to treatment. This study will assess the adverse events and how pivekimab sunirine moves through the body in pediatric participants with relapsed or refractory (R/R) AML.

Pivekimab sunirine is a drug being evaluated in the treatment of AML. This is an open label, single arm study, participants will be enrolled in 1 of the 3 cohorts based on their age and will receive pivekimab sunirine at a dose based on their weight. Around 18 pediatric participants with a diagnosis of AML will be enrolled in the study at approximately 30 sites around the world.

Participants will receive intravenous (IV) pivekimab sunirine alone. The total study duration is approximately 28 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed acute myeloid leukemia (AML) meeting one of the following disease criteria:

  * Second or greater relapse. OR
  * Disease refractory to second or subsequent line of therapy (defined as resistant disease after at least one cycle of each treatment regimen).
* Must have myeloid leukemic blasts that are CD123-positive by flow cytometry as determined by the treating institution.
* Has >= 5% myeloid leukemic blasts in bone marrow at time of relapse or refractory disease and prior to Screening for this study.
* Performance status by Lansky (< 16 years old at evaluation) or Karnofsky (>= 16 years old at evaluation) score >= 50 or ECOG score <= 2.
* May have status of central nervous system (CNS)1, CNS2, or CNS3 disease without clinical signs or neurologic symptoms suggestive of CNS leukemia, such as facial nerve palsy, brain/eye involvement or hypothalamic syndrome. Participants may have non-CNS extramedullary disease.
* For those participants who have not reached the age of consent, parent or legal guardian with the willingness and ability to provide informed consent and participant willing and able to give assent, as appropriate for age and country.

Exclusion Criteria:

* Known clinically significant cardiac disease.
* Down syndrome.
* Acute promyelocytic leukemia (APL) or juvenile myelomonocytic leukemia (JMML).
* Symptomatic central nervous system (CNS3) disease
* Prior history of any severity veno-occlusive disease/sinusoidal obstructive syndrome (VOD/SOS) of the liver.
* Prior history of hematopoietic stem cell transplant within 6 months prior to Screening.
* Have received prior Chimeric Antigen Receptor T-cell (CAR-T) therapy.
* Any other known current malignancy requiring therapy.
* Currently receiving anticancer therapy with antineoplastic intent, including radiotherapy, systemic therapy small molecules, monoclonal antibodies, other investigational agents, or high-dose chemotherapy with the exception of intrathecal therapy.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) Leading to Treatment Discontinuation | Up to Approximately 24 Months
  Number of participants with protocol specified Treatment-Emergent Adverse Events (TEAEs) during and after treatment with pivekimab sunirine (PVEK). Severity of TEAEs will be graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Maximum Observed Serum/Plasma Concentration (Cmax) of Intact Antibody-Drug Conjugate (ADC) | Up to Approximately 22 Months
  Maximum observed serum/plasma concentration of intact ADC.
Cmax of FGN849 Payload | Up to Approximately 22 Months
  Maximum observed serum/plasma concentration of FGN849 payload.
Area Under the Concentration-Time Curve (AUC) of Intact ADC | Up to Approximately 22 Months
  Area under the concentration-time curve of intact ADC.
AUC of FGN849 payload | Up to Approximately 22 Months
  Area under the concentration-time curve of FGN849 payload.
Time to Cmax (Tmax) of Intact ADC | Up to Approximately 22 Months
  Time to Cmax of intact ADC.
Tmax of FGN849 Payload | Up to Approximately 22 Months
  Time to Cmax of payload.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Complete Remission (CR) | Up to Approximately 28 Months
  CR is defined as Hematologic recovery: Absolute Neutrophil Count (ANC) >= 1.0 × 10^9/L (>= 1,000/μL) and platelet count >= 100 × 10^9/L (≥ 100,000/μL); < 5% bone marrow blasts; absence of circulating blasts; no evidence of extramedullary disease; no transfusions or support by exogenous growth factors (GCSF) within 7 days prior to response evaluation.
Percentage of Participants Achieving Composite Complete Remission (CR + complete remission with incomplete recovery [CRi]) | Up to Approximately 28 Months
  Percentage of participants achieving CR + CRi.
Percentage of Participants Achieving Composite Complete Remission (CR + complete remission with partial hematological [CRh]) | Up to Approximately 28 Months
  Percentage of participants achieving CR + CRh.
Duration of Complete Remission (DOCR) | Up to Approximately 28 Months
  DOCR is defined as the first response of CR to the time of relapse or death from any cause, whichever comes first; for participants who did not relapse or die, the duration will be censored at the time of the last response assessment.
Duration of Composite Complete Remission (CR + CRi) | Up to Approximately 28 Months
  Duration of composite complete remission (CR + CRi).
Duration of Composite Complete Remission (CR + CRh) | Up to Approximately 28 Months
  Duration of composite complete remission (CR + CRh).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-692